CLINICAL TRIAL: NCT00240409
Title: A Randomized Single-blind Placebo Controlled Comparative Trial of Pramipexole Tablets and Bromocriptine Tablets in Patients With Parkinson's Disease.
Brief Title: Randomized Single-blind Placebo Controlled Comparative Trial of Pramipexole and Bromocriptine in Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248.516
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole; Bromocriptine

INTERVENTIONS:
Drug: Pramipexole
Drug: Bromocriptine

SUMMARY:
The objective of this study was to investigate the efficacy and safety of Pramipexole Tablets in patients with Parkinson's disease (who can be treated with L-DOPA concomitantly) in a single blind, comparative method using Bromocriptine tablets as comparators (phase III comparative trial)

DETAILED DESCRIPTION:
The trial was to investigate the efficacy and safety of Pramipexole in patients with Parkinson's disease who can be concomitantly treated with L-DOPA in a double-blindmethod using Bromocriptine tablets as comparators (phase III comparative trial).

For efficacy evaluation, two primary endpoints were chosen:

* Totalled score according to Part III of UPDRS (motor examination)
* Totalled score according to Part II of UPDRS (activities of daily living)

The safety profile of the study drug was evaluated by physical examination, blood pressure, Electrocardiogram, Laboratory tests, AEs and SAEs.

Patients eligible for the trial who met all inclusion and exclusion criteria and who gave their informed consent were randomized to one of two treatment groups, i.e., Pramipexole tablets or Bromocriptine tablets. Patients were administered the study drug according to the dosing schedule.

The treatment period lasted maximal 12 weeks (ascending dose interval: up to 8 weeks, maintenance dose interval: 4 weeks or longer). In addition, a descending dose interval was 1-4 weeks.

Each patient received 7 visits except the patients drops or withdrawals:

visit 1: screening visit 2: randomization and baseline visit 3-6: ascending dose interval visit 7: Maintenance dose interval

Study Hypothesis:

Primary variables are both total of UPDRS (Unified Parkinson's Disease Rating Scale) part III items and of UPDRS part II items in change from baseline. The trial hypothesis is to demonstrate non-inferiority to Bromocriptine over an equivalence margin(=delta; the clinically largest difference judged as clinically acceptable) with 90% power, one sided for the above two primary variables at the error probability of 2.5% each. The equivalency margin for the primary variables (total of UPDRS Part III, and of UPDRS Part II) can be determined as 2.0 and 1.0 respectively referring to the results of oversea pivotal study of Pramipexole (BI Trial No. 248.326; U96-0232) and judged by the study investigator.

Comparison(s):

The primary endpoint of the study was the change of totalled score according to Part III of UPDRS (motor examination) and totalled score according to Part II of UPDRS (activities of daily living) after 12 weeks treatment of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-80 years
* Patients with idiopathic Parkinson's disease corresponding to stages II-IV according to the classification of Hoehn and Yahr during an "on" period, and/or patients in whom the individual optimized dosage of levodopa (and decarboxylase inhibitor) causes motor fluctuations characterized as end-of-dose phenomena or "wearing-off" effects for at least 30 days prior to initial administration of study medication and whose daily total "off" time is at least 2 hours and no more than 6 hours during waking time.
* Patients able to keep an accurate patient diary of the times of "on"- and "off"-periods during waking hours. Family members, guardians or nursing personnel may assist the patient.
* Informed Consent (consent in writing)

Exclusion Criteria:

* Patients with atypical parkinsonian syndromes due to drugs, metabolic disorders , encephalitis, or degenerative disease.
* Dementia that could impair compliance with medication, impair maintenance of accurate patient diaries, and/or preclude the signing of informed consent.
* History of psychosis except that which was elicited by treatment with levodopa or dopamine agonists unless the patient remains psychotic and in the opinion of the investigator would be unable to participate in the study.
* History of active epilepsy within the last two years prior to Visit 2.
* Patients with second or third degree AV block or sick sinus syndrome.
* Patients with resting heart rate below 50 beats per minute.
* Patients with congestive heart failure classified as functional Class III or IV by the New York Heart Association.
* Patients with myocardial infarction within six months of randomization.
* Patients with other clinical significant heart conditions which would negatively impact on the patient completing the study.
* Clinically significant kidney disease which may prevent the patient from completing the study and/or an elevation in either blood creatinine or urea nitrogen >1.5 times the laboratory normal.
* Clinically significant liver disease which may prevent the patient from completing the study and/or an elevation in either total bilirubin, SGPT, or SGOT of >1.5 times the laboratory normal.
* Retinopathia pigmentosa
* Presence of active neoplastic disease
* Patients with surgery within 180 days of Visit 2 which in the opinion of the investigator would negatively impact on the patient's participation in the clinical study or a history of stereotaxic brain surgery.
* At screening supine systolic blood pressure less than 100mmHg or evidence of a 20 mmHg decline in systolic blood pressure at one minute after standing compared with the previous supine systolic blood pressure obtained after 5 minutes of quiet rest in the supine position if the decline in blood pressure upon standing is associated with symptoms. Blood pressure at study entry (supine and standing) is expressed as the average of the second and third measured values.
* Patients who have received any of the following drugs during the 30 days prior to administered of study medication unless a longer period of time is specifically noted: neuroleptics (60 days), a-methyl-dopa, metoclopramide (60 days), flunarizine, cinnarizine, parenteral ergot preparation, bromocriptine, pergolide, A monoamine oxidase (MAO) inhibitors excluding l-deprenyl, methylphenidate hydrochloride, amphetamine derivatives, beta blockers (e.g. propranolol) only if used as an adjunctive treatment for PD, or reserpine.
* Females of childbearing potential not using oral contraceptives or a medically recognized mechanical means of contraception.
* Electroconvulsive therapy within 90 days of Visit 2.
* Patients who are participating in other drug studies or who receive other investigational drugs within 30 days prior to Visit 2, nor the patients previously randomized into this study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2003-07; Primary Completion 2004-08 (Actual); Study Completion 2004-08

PRIMARY OUTCOMES:
Totalled score according to Part III of UPDRS (motor examination) Totalled score according to Part II of UPDRS (activities of daily living)

SECONDARY OUTCOMES:
Totalled score of UPDRS Part IV, UPDRS Part I, the Modified Hoehn and Yahr Staging, Parkinson Dyskinesia Scale, and patient records.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (7):
- China (7):
  - First Hospital of Beijing University, Beijing
  - Beijing Tian Tan Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - General Hospital of PLA, Beijing
  - Shanghai Rui Jin Hospital, Shanghai
  - Hua Shan Hospital, Fu Dan University, Shanghai